CLINICAL TRIAL: NCT03646331
Title: A Phase I, Open-label, Randomised, Single-centre, 2-way Crossover Bioequivalence Study Comparing 2 Formulations of Imeglimin After Single Oral Doses in Healthy Caucasian Subjects
Brief Title: Bioequivalence of Imeglimin Tablet Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PXL008-022
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Bioequivalence
MeSH Terms: interventions — imeglimin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet A in Session 1 and Tablet B in Session 2 (Experimental): Tablet A = reference product Tablet B = test product
  Interventions: Drug: Imeglimin Reference product; Drug: Imeglimin
- Tablet B in Session 1 and Tablet A in Session 2 (Experimental): Tablet A = reference product Tablet B = test product
  Interventions: Drug: Imeglimin Reference product; Drug: Imeglimin

INTERVENTIONS:
Drug: Imeglimin Reference product — Reference product
Drug: Imeglimin — Test product (new formulation tablet)

SUMMARY:
This is an open-label assessment of the bioequivalence of two 500 mg-tablet formulations of imeglimin (Tablet A [reference product] and Tablet B [test product]), in at least 16 healthy Caucasian volunteers.

ELIGIBILITY:
Inclusion Criteria:

* BMI : 18.5-29.9
* Body weight ≥ 60 kg
* willing to use reliable contraception
* able to give fully informed written consent.

Exclusion Criteria:

* Positive tests for hepatitis B & C, HIV
* severe adverse reaction to any drug; sensitivity to trial medication and/or food allergies
* drug or alcohol abuse
* smoking of more than 5 cigarettes daily or drinking more than 5 cups of caffeinated drinks daily
* over-the-counter medication, vitamins and herbal remedies, or prescribed medication in the 20 days before the first dose of trial medication (with the exception of paracetamol [acetaminophen] and oral contraception);
* participation in other clinical trials of unlicensed medicines, or loss of more than 400 mL blood, within the previous 3 months
* vital signs outside the acceptable range
* clinically relevant abnormal findings at the screening assessment; estimated glomerular filtration rate (eGFR) at screening < 80 mL/min/1.73 m2
* acute or chronic illness
* clinically relevant abnormal medical history or concurrent medical condition;
* surgery or medical condition that might affect the absorption of medicines;
* possibility that volunteer will not cooperate
* pre-menopausal females who are pregnant or lactating, or who are sexually active and not using a reliable method of contraception;
* objection by the volunteer's General Practitioner (GP).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Pk parameters of imeglimin | from dosing up to 48h
  Cmax: peak plasma concentration after dosing

SECONDARY OUTCOMES:
PK parameters of Imeglimin | from dosing up to 48h
  AUC last: area Under the concentration time curve
Incidence of treatment emergent adverse events (Safety and tolerability) | From Day 1 to Day 15
  Incidence of treatment emergent adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom